CLINICAL TRIAL: NCT01593930
Title: Evaluation of the Success Rate of Pulpal Anesthesia in Mandibular First Molar Following Infiltration of 4% Articaine Alone and as Supplemental Injection After Inferior Alveolar Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahedan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Kaveh Oloomi, DDS, MS, Assistant Professor, Zahedan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Articaine pulpal anesthesia
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Pulpal Anesthesia
Keywords: Pulp Anesthesia; Articaine; Lidocaine
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 Articaine(Infiltration) (Experimental): Buccal infiltration of one 4% Articaine cartridge with 1/100000 epinephrine
  Interventions: Other: 1 Articaine(Infiltration)
- 2 Articaine(Infiltration) (Experimental): Buccal infiltration of two 4% Articaine cartridges with 1/100000 epinephrine
  Interventions: Other: 2 Articaine(Infiltration)
- Lidocaine(IANB)+1Articaine(Infiltration) (Experimental): Inferior alveolar nerve block using one 2% Lidocaine cartridge with 1/80000 epinephrine + Buccal infiltration of one 4% Articaine cartridge with 1/100000 epinephrine
  Interventions: Other: Lidocaine(IANB)+1Articaine(Infiltration)
- Lidocaine(IANB) (Experimental): Inferior alveolar nerve block using one 2% Lidocaine cartridge with 1/80000 epinephrine
  Interventions: Other: Lidocaine(IANB)

INTERVENTIONS:
Other: Lidocaine(IANB) — Inferior alveolar nerve block using one 2% Lidocaine cartridge with 1/80000 epinephrine
  Other Names: Persocaine E
  Arms: Lidocaine(IANB)
Other: 1 Articaine(Infiltration) — Buccal infiltration of one 4% Articaine cartridge with 1/100000 epinephrine
  Other Names: Septanest
  Arms: 1 Articaine(Infiltration)
Other: 2 Articaine(Infiltration) — Buccal infiltration of two 4% Articaine cartridges with 1/100000 epinephrine
  Other Names: Septanest
  Arms: 2 Articaine(Infiltration)
Other: Lidocaine(IANB)+1Articaine(Infiltration) — Inferior alveolar nerve block using one 2% Lidocaine cartridge with 1/80000 epinephrine + Buccal infiltration of one 4% Articaine cartridge with 1/100000 epinephrine
  Other Names: Persocaine E + Septanest
  Arms: Lidocaine(IANB)+1Articaine(Infiltration)

SUMMARY:
The purpose of this study is to determine the success rate of pulpal anesthesia in mandibular firs molar following infiltration of 4% articaine alone and as supplemental injection after inferior alveolar nerve block(IANB).

DETAILED DESCRIPTION:
According to inclusion & exclusion criteria, volunteers will be selected and divided into 4 groups randomly. The clinician who does the injections will not be aware of study purpose. Also the person who does the electric pulp test (EPT); the volunteer and the statistical analyzer will not be aware of group codes. Intervention in each group will be as follow: Group 1-Buccal infiltration of one 4% Articaine cartridge with 1/100000 epinephrine. Group 2-Buccal infiltration of two 4% Articaine cartridges with 1/100000epinephrine. Group 3-Inferior alveolar nerve block using one 2% Lidocaine cartridge with 1/80000 epinephrine + buccal infiltration of one 4% Articaine cartridge with 1/100000 epinephrine. Group 4- Inferior alveolar nerve block using one 2% Lidocaine cartridge with 1/80000 epinephrine. Before injection a control tooth (contralateral canine) will be tested to understand the accuracy of patient's response to EPT; also for measuring the base line vitality, each tooth will be evaluated by EPT twice before injection. After injection each tooth will be evaluated by EPT every 3 minutes; also every minute the anesthesia of lip and tongue will be checked, up to 15 minutes. The tooth will be discerned "anesthetized" if the subject will not response to 80 reading of EPT in 2 consecutive tests. Finally the information will be recorded and in addition to the success rate the mean time for onset of anesthesia and its mean duration time will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 1 vital first mandibular molar without any restoration or decay

Exclusion Criteria:

* Patients with systemic conditions which eliminate the use of epinephrine
* Patients with history of allergy to amide anesthetics or contents of local anesthetic cartridge
* Pregnant women
* Use of analgesics, opioids or any other drugs which influence the anesthesia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Success rate | Every 3 minutes after injection
  Changes in tooth response to Electric Pulp Tester (EPT) will be checked each 3 minutes after injection. The anesthesia will be considered successful if the subject will not response to EPT at the 80 reading in 2 consecutive tests.

SECONDARY OUTCOMES:
Onset of anesthesia | Every 3 minutes after injection
  Changes in tooth response to Electric Pulp Tester (EPT) will be checked each 3 minutes after injection. No response from the patient at the 80 reading of EPT in 2 consecutive tests will be discerned as "completely anesthetized" and the time will be recorded as "onset of anesthesia".
Duration of anesthesia | Every 3 minutes after onset of anesthesia
  Changes in tooth response to Electric Pulp Tester (EPT) will be checked each 3 minutes after onset of anesthesia to determine when the subject will response again at the 80 reading of EPT.

CONTACTS AND LOCATIONS:
Overall Officials: Kaveh Oloomi, DDS, MS, Principal Investigator — Assistant Professor
Locations (1):
- Zahedan university of medical sciences, Vice-chancellor for research, Zahedan, Iran